CLINICAL TRIAL: NCT04886583
Title: Preliminary Multi-centric Clinical Study Assessing the Accuracy of the Non-invasive Wireless Armband Gabi Baby Band for the Continuous Monitoring and Recording of Vital Physiological Parameters on Infants and Young Children by Comparison of Simultaneous Polysomnographic Recording During Standard of Care Hospitalisation
Brief Title: Assessment of the Accuracy of the Non-invasive Wireless Armband Gabi Baby Band for Continuous Vital Parameters Monitoring in Infants and Young Children
Acronym: WAGSC1
Status: Completed | Type: Observational
Sponsor: Gabi SmartCare (Industry)
Responsible Party: Sponsor
Other Study IDs: WAGSC1
Record Dates: First submitted 2021-05-03; First posted 2021-05-14 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Blood Oxygen Desaturations; Sleep-Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gabi Baby Band: GSC 1
  Interventions: Device: Gabi Baby Band

INTERVENTIONS:
Device: Gabi Baby Band — Every enrolled patient must wear the Gaby Baby Band on the left arm in the aim to perform data analytics after the test has been performed

SUMMARY:
During a polysomnography test (PSG) previously prescribed by a physician, the patient also wears the Gaby Baby Band (GBB) during an entire night of sleep. After the test, data from the device and from the PSG (HR, SpO2, BR) will be saved and analysed in the aim to assess the actual accuracy of the GBB with golden standard values (ECG, Oximeter, belly belt). In a second analysis, the aim is to improve the accuracy of the GBB algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children under 5 years of age
* PSG is required per standard of care
* Signature of consent form

Exclusion Criteria:

* Children having already done the PSG wearing GBB for this study
* Epileptic children (due to high motion/artifacts during sleep)
* Weight below 2.5 kg

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children under 5 years old who need to undergo a polysomnographic exam, as per standard of care, and admitted in the PSG paediatrics service for at least 1 night after proper medical examination and diagnostic by a qualified physician.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
to improve the calibration, the correctness and reproducibility of the SpO2 (%) measurements reported by the GBB | 12 hours
  The primary objective of this pilot study is to improve the calibration, the correctness and reproducibility of the measurements reported by the GBB compared to a standard of care for measuring SpO2 (%) through the recording of raw data with the Gabi Baby Band in parallel with values recorded by medical devices used by the investigation site in its current standard care practice test (during sleep) on infants and children under 5 years old.

SECONDARY OUTCOMES:
to improve the calibration, the correctness and reproducibility of the measurements of the BR (breathing rate; cycle/min) reported by the GBB | 12 hours
  The primary objective of this pilot study is to improve the calibration, the correctness and reproducibility of the measurements reported by the GBB compared to a standard of care for measuring BR (breathing rate; cycle/min) through the recording of raw data with the Gabi Baby Band in parallel with values recorded by medical devices used by the investigation site in its current standard care practice test (during sleep) on infants and children under 5 years old.
to improve the calibration, the correctness and reproducibility of the measurements of the HR (heart rate; beat/min or bpm) reported by the GBB | 12 hours
  The primary objective of this pilot study is to improve the calibration, the correctness and reproducibility of the measurements reported by the GBB compared to a standard of care for measuring BR (heart rate; beat/min) through the recording of raw data with the Gabi Baby Band in parallel with values recorded by medical devices used by the investigation site in its current standard care practice test (during sleep) on infants and children under 5 years old.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Hopital Universitaire Des Enfants Reine Fabiola, Jette, Brussels Capital
  - CHU Marie Curie, Charleroi, Hainaut
  - CHC Montlégia, Liège

IPD SHARING:
Plan to Share IPD: Undecided